CLINICAL TRIAL: NCT05111249
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Range Finding Study With Open-Label Extension to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of LMI070/Branaplam Administered as Weekly Oral Doses in Participants With Early Manifest Huntington's Disease
Brief Title: A Dose Range Finding Study With Open-Label Extension to Evaluate the Safety of Oral LMI070/Branaplam in Early Manifest Huntington's Disease
Acronym: VIBRANT-HD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was halted prematurely due to signs and symptoms that suggested the possibility of peripheral neuropathy. All participants who received branaplam continued to undergo routine (safety) evaluations for up to a year following their final dose
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLMI070C12203; 2020-000105-92 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Early Manifest Huntington Disease
Keywords: Early Manifest; Huntington Disease; Branaplam; LMI070; Dose Range Finding; Safety; HD; mHTT; Pharmacokinetics; oral; Adult
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: The study design used a staggered cohort approach, allowing safety and tolerability of lower doses to be assessed before randomizing subjects to higher doses.
  At the time of the Cohort Gating Assessments (CGAs), all available data was reviewed from a safety and dose finding perspective by an independent Sponsor team to support the decision to open the next cohort. The independent Data Monitoring Committee (DMC) reviewed the data separately. The decision to open a new cohort was planned to be made by the Sponsor in consultation with the DMC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This was a randomized double blind study. Participants were planned to be randomized in an equal randomization rate among the open treatment arms, and then in a 4:1 ratio for active vs. placebo within each arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Arm A (Experimental): Branaplam 56 mg oral solution once weekly
  Interventions: Drug: Branaplam
- Treatment Arm B (Experimental): Branaplam 112 mg oral solution once weekly
  Interventions: Drug: Branaplam
- Treatment Arm C or X or Y (Experimental): (C) Branaplam 154 mg oral solution once weekly, OR (X) Branaplam 84 mg oral solution once weekly OR (Y) Branaplam 28 mg oral solution once weekly
  Interventions: Drug: Branaplam
- Placebo (Placebo Comparator): Matching placebo oral solution once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branaplam — messenger ribonucleic acid (RNA) splicing modifier. Branaplam was administered as an oral solution once weekly.
  Other Names: LMI070
  Arms: Treatment Arm A; Treatment Arm B; Treatment Arm C or X or Y
Drug: Placebo — Matching placebo oral solution once weekly
  Arms: Placebo

SUMMARY:
This is the first study of branaplam in adults with Huntington's Disease (HD) to determine the correct dose required to lower mutant huntingtin protein (mHTT) levels in the cerebrospinal fluid (CSF) to a degree expected to be efficacious over longer periods of time.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled study with a variable duration (between approximately 17 weeks to approximately 53 weeks) for the core period and a one-year open label extension (OLE) in early-stage manifest Huntington's disease (HD) participants.

After screening period and baseline assessments, the following two Treatment Periods were planned:

• The core period consisted of a 17-week double-blind, placebo-controlled, Dose Range Finding (DRF) portion of the study, followed by a blinded extension (BE) of variable duration (up to approximately 53 weeks). The DRF Period was to evaluate the safety, tolerability, pharmacokinetivs (PK) and pharmacodynamics (PD) of branaplam, as well as determine the optimal dose(s) to explore in further clinical evaluations.

The core period was planned to consist of 3 treatment arms:

* Cohort 1: Treatment Arm A: branaplam 56 mg oral solution or matching placebo, once weekly
* Cohort 2: Treatment Arm B: branaplam 112 mg oral solution or matching placebo, once weekly
* Cohort 3:

Treatment Arm C: branaplam 154 mg oral solution or matching placebo, once weekly or Treatment Arm X: branaplam 84 mg oral solution or matching placebo, once weekly or Treatment Arm Y: branaplam 28 mg oral solution or matching placebo, once weekly

• The OLE was a one-year open-label extension to assess both long-term safety and tolerability, as well as the efficacy of the recommended optimal dose(s) for branaplam.

Due to safety concerns an urgent safety measure (USM) follow-up notification dated 06-Dec-2022 was issued to permanently discontinue the study treatment in all participants. At that point, only cohort 1 was enrolled. Therefore, only cohort 1 data is available for analysis (Treatment Arm A: branaplam 56 mg oral solution or matching placebo, once weekly). Participants who received active treatment (branaplam) were to remain in the study for follow-up for approximately one year following initial treatment discontinuation. The OLE part was not opened.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent must be obtained prior to participation in the study.
* Clinically diagnosed Stage 1 or 2 Huntington's disease with a diagnostic confidence level (DCL) = 4 and a United Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity (TFC) >8 at screening.
* Genetically confirmed Huntington's disease, with presence of ≥40 cytosine-adenineguanine (CAG) repeats in the huntingtin gene.
* Male and female participants between 25 to 75 years of age, inclusive, on the day of Informed Consent signature.

Exclusion Criteria

* Prior participation in clinical trial investigating a huntingtin-lowering therapy (unless participant received only placebo).
* Participants taking medications prohibited by the protocol.
* Any medical history, lumbar surgery or condition that would interfere with the ability to complete the protocol specified assessments.
* Participant has other severe, acute or chronic medical conditions including unstable psychiatric conditions, or laboratory abnormalities that in the opinion of the Investigator may increase the risk associated with study participation, or that may interfere with the interpretation of the study results.
* Any surgical or medical condition which might put the participant at risk in case of participation in the study. The Investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence at the Screening visit.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (3):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
- Germany (3):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Borowsky B, Ramos H, Caputo A, Hartmann A, Faller T, Peters T, Sui Y, Liu F, Meadowcroft M, David OJ, Laisney M, Kinhikar A, Marder KS, Tabrizi SJ, Landwehrmeyer GB, Leavitt BR. Oral splicing modulator branaplam in Huntington's disease: a phase 2 randomized controlled trial. Nat Med. 2026 Jan;32(1):103-112. doi: 10.1038/s41591-025-04117-4. Epub 2026 Jan 5. PMID 41491108
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: March 2024. J Huntingtons Dis. 2024;13(1):1-14. doi: 10.3233/JHD-240017. PMID 38489195
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: November 2022. J Huntingtons Dis. 2022;11(4):351-367. doi: 10.3233/JHD-229006. PMID 36463457
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 12 investigative sites in 5 countries.
Pre-assignment Details: The Screening period had a duration of up to 6 weeks. For eligible participants, the baseline measurements were performed within 6 days prior to the first dose of study treatment. At the Week 1 visit in the Core period participants were randomized (4:1) to receive either branaplam or placebo.
  The last study visit was performed at Week 69. The open label extension (OLE) period was not opened.
Groups:
- Placebo: Treatment Arm A: matching placebo oral solution once weekly
- Branaplam 56 mg: Treatment Arm A: branaplam 56 mg oral solution once weekly
Period: Overall Study
Arm/Group | Placebo | Branaplam 56 mg
Started | 5 | 21
Completed | 4 | 13
Not Completed | 1 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Participant decision | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Branaplam 56 mg | Total
Number analyzed (Participants) | 5 | 21 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.30) | 49.6 (10.06) | 50.2 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 11
  Male | 4 | 11 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 18 | 23
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to Week 17 in mHTT Protein in CSF
Description: Mutant Huntingtin (mHTT) protein was measured in cerebrospinal fluid (CSF) obtained via lumbar puncture. The percentage change from baseline to Week 17 in mHTT protein in CSF was calculated with the following formula: (mHTTweek17 - mHTTbaseline)/ mHTTbaseline * 100.
  Baseline value for mHTT is the last evaluable measurements prior to the first administration of study drug.
Time Frame: Baseline, Week 17
Population: Participants in the Safety Analysis Set (SAF) who had an available value for the outcome measure at baseline and Week 17. SAF included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: % change in mHTT protein
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 4 | 9
% change in mHTT protein | -1.38 (20.517) | -26.61 (22.354)

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence of AEs (any AEs regardless of seriousness) and SAEs, including changes in vital signs, neurological examination, electrocardiograms (ECGs) and laboratory parameters qualifying and reported as AEs.
  Participants received study treatment up to maximum Week 20 (placebo) and Week 22 (branaplam).
Time Frame: From first dose of study treatment up to Week 69
Population: Safety Analysis Set including all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 21
Participants
  AEs | 2 | 18
  Study drug-related AEs | 1 | 14
  SAEs | 0 | 4
  Study drug-related SAEs | 0 | 3

3. Secondary Outcome: Percentage Change From Baseline in Total Brain Volume
Description: Three-dimensional magnetic resonance imaging (MRI) data was acquired and used to measure brain volume at each time point and changes in brain volume longitudinally. Brain MRI scans were performed at each time point without gadolinium contrast.
  Changes in volumetric MRI were measured in regions of interests: ventricular, caudate (left and right) and total brain volume.
  The baseline MRI scan was obtained within 6 days prior to the first dose of study treatment.
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: Participants in the Safety Analysis Set (SAF) who had an available value for the outcome measure at baseline and the corresponding study visit. SAF included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: % change in total brain volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 4 | 17
% change in total brain volume
  Week 17 | -0.20 (0.332) | -0.43 (2.362)
  Week 33: number analyzed (Participants) | 3 | 17
  Week 33 | -0.67 (0.352) | -0.88 (0.681)
  Week 53: number analyzed (Participants) | 1 | 12
  Week 53 | -0.25 | -1.34 (0.848)
  Week 69: number analyzed (Participants) | 0 | 12
  Week 69 |  | -1.63 (0.877)

4. Secondary Outcome: Percentage Change From Baseline in Total Brain Volume Excluding Patients With Subdural Hematoma
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: Participants in the Safety Analysis Set (SAF) who had an available value for the outcome measure at baseline and the corresponding study visit, and who did not have subdural hematoma. SAF included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: % change in total brain volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 4 | 15
% change in total brain volume
  Week 17 | -0.20 (0.332) | -1.09 (0.599)
  Week 33: number analyzed (Participants) | 3 | 15
  Week 33 | -0.67 (0.352) | -0.80 (0.675)
  Week 53: number analyzed (Participants) | 1 | 10
  Week 53 | -0.25 | -1.30 (0.748)
  Week 69: number analyzed (Participants) | 0 | 10
  Week 69 |  | -1.68 (0.751)

5. Secondary Outcome: Percentage Change From Baseline in Lateral Ventricles Volume
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % change in lateral ventricles volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 3 | 17
% change in lateral ventricles volume
  Week 17 | 1.63 (1.392) | 8.84 (11.599)
  Week 33 | 5.51 (1.772) | 11.73 (9.799)
  Week 53: number analyzed (Participants) | 1 | 12
  Week 53 | 3.43 | 15.77 (10.842)
  Week 69: number analyzed (Participants) | 0 | 12
  Week 69 |  | 17.40 (10.182)

6. Secondary Outcome: Percentage Change From Baseline in Lateral Ventricles Volume Excluding Patients With Subdural Hematoma
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change in lateral ventricles volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 3 | 15
% change in lateral ventricles volume
  Week 17 | 1.63 (1.392) | 9.47 (6.061)
  Week 33 | 5.51 (1.772) | 9.43 (5.673)
  Week 53: number analyzed (Participants) | 1 | 10
  Week 53 | 3.43 | 12.38 (6.193)
  Week 69: number analyzed (Participants) | 0 | 10
  Week 69 |  | 14.45 (6.040)

7. Secondary Outcome: Percentage Change From Baseline in Left Caudate Volume
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % change in left caudate volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 4 | 17
% change in left caudate volume
  Week 17: number analyzed (Participants) | 4 | 16
  Week 17 | -0.93 (3.782) | -4.44 (3.005)
  Week 33: number analyzed (Participants) | 3 | 17
  Week 33 | -3.95 (2.147) | -4.30 (3.331)
  Week 53: number analyzed (Participants) | 1 | 11
  Week 53 | -2.69 | -6.33 (4.417)
  Week 69: number analyzed (Participants) | 0 | 12
  Week 69 |  | -5.44 (7.864)

8. Secondary Outcome: Percentage Change From Baseline in Left Caudate Volume Excluding Patients With Subdural Hematoma
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change in left caudate volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 4 | 15
% change in left caudate volume
  Week 17: number analyzed (Participants) | 4 | 14
  Week 17 | -0.93 (3.782) | -4.14 (2.300)
  Week 33: number analyzed (Participants) | 3 | 15
  Week 33 | -3.95 (2.147) | -3.58 (2.692)
  Week 53: number analyzed (Participants) | 1 | 9
  Week 53 | -2.69 | -6.24 (4.788)
  Week 69: number analyzed (Participants) | 0 | 10
  Week 69 |  | -4.81 (8.351)

9. Secondary Outcome: Percentage Change From Baseline in Right Caudate Volume
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % change in right caudate volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 3 | 17
% change in right caudate volume
  Week 17 | -3.28 (3.496) | -2.79 (4.604)
  Week 33 | -6.91 (1.895) | -4.11 (4.146)
  Week 53: number analyzed (Participants) | 1 | 11
  Week 53 | -5.34 | -6.81 (4.251)
  Week 69: number analyzed (Participants) | 0 | 12
  Week 69 |  | -6.34 (6.934)

10. Secondary Outcome: Percentage Change From Baseline in Right Caudate Volume Excluding Patients With Subdural Hematoma
Description: as for outcome 3
Time Frame: Baseline, Week 17, Week 33, Week 53, Week 69
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change in right caudate volume
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 3 | 15
% change in right caudate volume
  Week 17 | -3.28 (3.496) | -2.67 (4.850)
  Week 33 | -6.91 (1.895) | -3.23 (3.437)
  Week 53: number analyzed (Participants) | 1 | 9
  Week 53 | -5.34 | -6.57 (4.418)
  Week 69: number analyzed (Participants) | 0 | 10
  Week 69 |  | -5.60 (7.249)

11. Secondary Outcome: Change From Baseline in the Unified Huntington's Disease Rating Scales (UHDRS) Total Functional Capacity (TFC)
Description: The TFC focuses on the investigator's assessment of the participant's capacity to perform a range of activities of daily living. The responses are derived from interview with the participant and/or companion, if applicable. TFC score range from 0 to 13, with higher scores representing better functioning.
Time Frame: Baseline, Week 17, Week 33 and Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 19
score on scale
  Week 17 | -1.0 (2.35) | -0.8 (2.39)
  Week 33: number analyzed (Participants) | 4 | 17
  Week 33 | -0.5 (2.52) | -1.3 (2.31)
  Week 69: number analyzed (Participants) | 0 | 13
  Week 69 |  | -1.2 (2.94)

12. Secondary Outcome: Change From Baseline in the Unified Huntington's Disease Rating Scales (UHDRS) Total Motor Scale (TMS)
Description: The TMS is the cumulative sum of the individual motor ratings obtained during the administration of the motor assessment portion of the UHDRS. TMS score range from 0 to 124 with higher scores representing more significant impairment.
Time Frame: Baseline, Week 17, Week 33 and Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 19
score on scale
  Week 17 | 6.0 (11.29) | 5.1 (9.14)
  Week 33: number analyzed (Participants) | 4 | 17
  Week 33 | 2.5 (10.34) | 2.6 (8.83)
  Week 69: number analyzed (Participants) | 0 | 13
  Week 69 |  | 3.6 (8.99)

13. Secondary Outcome: Change From Baseline in the Unified Huntington's Disease Rating Scales (UHDRS) Independence Scale (IS)
Description: The IS represents the investigator's assessment of the participant's level of independence, including topics of employment, finances, self-care and feeding. The scale has 19 discrete scores, from 10 (tube fed, total bed care) to 100 (no special care needed) with 5-point increments in between.
Time Frame: Baseline, Week 17, Week 33 and Week 69
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 19
score on scale
  Week 17 | -1.0 (11.40) | -1.8 (9.16)
  Week 33: number analyzed (Participants) | 4 | 17
  Week 33 | 1.3 (16.52) | -4.7 (8.19)
  Week 69: number analyzed (Participants) | 0 | 13
  Week 69 |  | -6.5 (13.29)

14. Secondary Outcome: Concentrations of mHTT Protein and Total HTT in CSF
Description: Mutant Huntingtin (mHTT) protein and total HTT measured in cerebrospinal fluid (CSF) obtained via lumbar puncture.
  Baseline value is the last evaluable measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 9, Week 17
Population: Participants in the Safety Analysis Set (SAF) who had an available value for the outcome measure at the corresponding study visit. SAF included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: fmol
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 21
fmol
  mHTT - Baseline | 86.14 (35.590) | 102.03 (48.533)
  mHTT - Week 9: number analyzed (Participants) | 5 | 17
  mHTT - Week 9 | 86.31 (43.265) | 74.68 (37.111)
  mHTT - Week 17: number analyzed (Participants) | 4 | 9
  mHTT - Week 17 | 77.68 (33.077) | 65.58 (41.152)
  Total HTT - Baseline | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF. | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF.
  Total HTT - Week 9 | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF. | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF.
  Total HTT - Week 17 | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF. | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in CSF.

15. Secondary Outcome: Concentrations of mHTT Protein and Total HTT in Plasma
Description: Mutant Huntingtin (mHTT) protein and total HTT measured in plasma. Baseline value is the last evaluable measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 17
Population: Safety Analysis Set (SAF)
Measure: Mean (Standard Deviation); unit: fmol
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 21
fmol
  mHTT - Baseline | NA (NA) — Assay issues did not allow a reliable quantification of mHTT protein in plasma. | NA (NA) — Assay issues did not allow a reliable quantification of mHTT protein in plasma.
  mHTT - Week 17 | NA (NA) — Assay issues did not allow a reliable quantification of mHTT protein in plasma. | NA (NA) — Assay issues did not allow a reliable quantification of mHTT protein in plasma.
  Total HTT - Baseline | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in plasma. | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in plasma.
  Total HTT - Week 17 | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in plasma. | NA (NA) — Assay issues did not allow a reliable quantification of total HTT in plasma.

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Branaplam and Its Metabolite UFB112
Description: Pharmacokinetic (PK) parameters were calculated based on branaplam and its metabolite UFB112 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: pre-dose and 4, 7, 12, 22, 72 and 168 hours after branaplam dose at Week 1 and Week 17
Population: Patients in the PK analysis set with an available value for the outcome measure at each timepoint. The PK Analysis Set is only applicable to patients treated with branaplam and includes all participants with at least one evaluable concentration data sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 21
ng/mL
  Branaplam - Week 1 | 26.1 (7.99)
  Branaplam - Week 17: number analyzed (Participants) | 4
  Branaplam - Week 17 | 45.3 (7.96)
  UFB112 - Week 1 | 31.9 (12.6)
  UFB112 - Week 17: number analyzed (Participants) | 4
  UFB112 - Week 17 | 53.3 (20.4)

17. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Branaplam and Its Metabolite UFB112
Description: PK parameters were calculated based on branaplam and its metabolite UFB112 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: pre-dose and 4, 7, 12, 22, 72 and 168 hours after branaplam dose at Week 1 and Week 17
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 21
hours
  Branaplam - Week 1 | 7.00 [3.77 to 23.0]
  Branaplam - Week 17: number analyzed (Participants) | 4
  Branaplam - Week 17 | 4.18 [4.00 to 7.00]
  UFB112 - Week 1 | 7.00 [4.00 to 72.00]
  UFB112 - Week 17: number analyzed (Participants) | 4
  UFB112 - Week 17 | 14.5 [4.28 to 22.00]

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 168 Hours (AUC0-168h) of Branaplam and Its Metabolite UFB112
Description: PK parameters were calculated based on branaplam and its metabolite UFB112 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-168h calculation.
Time Frame: pre-dose and 4, 7, 12, 22, 72 and 168 hours after branaplam dose at Week 1 and Week 17
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 21
hr*ng/mL
  Branaplam - Week 1: number analyzed (Participants) | 20
  Branaplam - Week 1 | 1880 (368)
  Branaplam - Week 17: number analyzed (Participants) | 4
  Branaplam - Week 17 | 3190 (455)
  UFB112 - Week 1 | 3670 (1560)
  UFB112 - Week 17: number analyzed (Participants) | 4
  UFB112 - Week 17 | 5640 (2750)

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Branaplam and Its Metabolite UFB112
Description: PK parameters were calculated based on branaplam and its metabolite UFB112 plasma concentrations by using non-compartmental methods. The linear trapezoidal method and the regression analysis of the terminal elimination phase were used for AUCinf calculation.
Time Frame: pre-dose and 4, 7, 12, 22, 72 and 168 hours after branaplam dose at Week 1
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 21
hr*ng/mL
  Branaplam - Week 1: number analyzed (Participants) | 13
  Branaplam - Week 1 | 2270 (467)
  UFB112 - Week 1: number analyzed (Participants) | 1
  UFB112 - Week 1 | 3530

20. Secondary Outcome: Trough Concentration (Ctrough) of Branaplam and Its Metabolite UFB112 in Plasma
Description: Branaplam and its metabolite UFB112 concentrations were determined in plasma. Ctrough is defined as the concentration reached immediately before the next dose is administered. All drug concentrations below the lower limit of quantification were treated as zero for the calculation of PK parameters.
Time Frame: pre-dose at Weeks 2, 3, 5, 9, 13 and 17
Population: Patients in the PK analysis set with an available value for the outcome measure at each timepoint. The PK Analysis Set is only applicable to patients treated with branaplam and included all participants with at least one evaluable concentration data sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 20
ng/mL
  Branaplam - Week 2 | 4.10 (1.29)
  Branaplam - Week 3 | 6.54 (1.78)
  Branaplam - Week 5 | 8.50 (3.20)
  Branaplam - Week 9: number analyzed (Participants) | 15
  Branaplam - Week 9 | 7.85 (2.12)
  Branaplam - Week 13: number analyzed (Participants) | 9
  Branaplam - Week 13 | 8.54 (2.27)
  Branaplam - Week 17: number analyzed (Participants) | 6
  Branaplam - Week 17 | 7.88 (2.11)
  UFB112 - Week 2 | 12.1 (6.22)
  UFB112 - Week 3 | 18.0 (8.25)
  UFB112 - Week 5 | 21.9 (11.5)
  UFB112 - Week 9: number analyzed (Participants) | 15
  UFB112 - Week 9 | 21.2 (11.5)
  UFB112 - Week 13: number analyzed (Participants) | 9
  UFB112 - Week 13 | 18.5 (8.71)
  UFB112 - Week 17: number analyzed (Participants) | 6
  UFB112 - Week 17 | 16.1 (5.33)

21. Secondary Outcome: Trough Concentration (Ctrough) of Branaplam and Its Metabolite UFB112 in CSF
Description: Branaplam and its metabolite UFB112 concentrations were determined in cerebrospinal fluid (CSF) obtained via lumbar puncture. Ctrough is defined as the concentration reached immediately before the next dose is administered. All drug concentrations below the lower limit of quantification were treated as zero for the calculation of PK parameters.
Time Frame: pre-dose at Weeks 9 and 17
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 12
ng/mL
  Branaplam - Week 9 | 0.870 (0.311)
  Branaplam - Week 17: number analyzed (Participants) | 5
  Branaplam - Week 17 | 0.602 (0.355)
  UFB112 - Week 9 | 0.269 (0.184)
  UFB112 - Week 17: number analyzed (Participants) | 5
  UFB112 - Week 17 | 0.230 (0.154)

22. Secondary Outcome: Concentration Ratio CSF/Plasma of Branaplam and Its Metabolite UFB112
Description: Branaplam and its metabolite UFB112 concentrations were determined plasma and in cerebrospinal fluid (CSF) obtained via lumbar puncture. Concentration ratios CSF/plasma were calculated for subjects for whom CSF and plasma concentrations were available at the respective time point.
Time Frame: pre-dose at Weeks 9 and 17
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: concentration ratio
Arm/Group | Branaplam 56 mg
Number analyzed (Participants) | 11
concentration ratio
  Branaplam - Week 9 | 0.115 (NA) — In alignment with the secondary endpoints defined in the protocol, the statistical analysis plan (SAP) included only the calculation of the mean concentration ratio CSF/plasma. Therefore, no dispersion values were derived.
  Branaplam - Week 17: number analyzed (Participants) | 4
  Branaplam - Week 17 | 0.0864 (NA) — In alignment with the secondary endpoints defined in the protocol, the statistical analysis plan (SAP) included only the calculation of the mean concentration ratio CSF/plasma. Therefore, no dispersion values were derived.
  UFB112 - Week 9 | 0.0141 (NA) — In alignment with the secondary endpoints defined in the protocol, the statistical analysis plan (SAP) included only the calculation of the mean concentration ratio CSF/plasma. Therefore, no dispersion values were derived.
  UFB112 - Week 17: number analyzed (Participants) | 4
  UFB112 - Week 17 | 0.0161 (NA) — In alignment with the secondary endpoints defined in the protocol, the statistical analysis plan (SAP) included only the calculation of the mean concentration ratio CSF/plasma. Therefore, no dispersion values were derived.

23. Other Pre Specified Outcome: Number of Participants With NfL Increase and Recovery
Description: Neurofilament light chain (NfL) is a neuronal cytoplasmic protein highly expressed in large calibre myelinated axons. Its levels increase in cerebrospinal fluid (CSF) and serum in case of axonal damage in a variety of neurological disorders.
  The levels of NfL were determined in serum and CSF and the following 3 categories were defined:
  * Serum NfL (sNfL) increase: > 100 pg/mL or > 2 x baseline (BL) sNfL
  * sNfL recovery: Worsening criteria are no longer met (sNfL <= 100 pg/mL or sNfL <= 2 x BL sNfL) for visits after last visit with increase
  * CSF NfL increase: > 10000 pg/mL or > 2 x BL CSF NfL or > 2 x CSF NfL of the previous assessment
Time Frame: From baseline (before first dose of study treatment) up to Week 17 (CSF) and Week 69 (serum)
Population: Safety Analysis Set including all participants who received at least one dose of study drug. sNfL recovery was assessed in participants meeting the criterion for sNfL increase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Branaplam 56 mg
Number analyzed (Participants) | 5 | 21
Participants
  sNfL increase | 0 | 16
  sNfL recovery: number analyzed (Participants) | 0 | 16
  sNfL recovery | 0 | 14
  CSF NfL increase | 0 | 13

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to Week 69
Groups:
- Overall: All participants
Arm/Group | Placebo | Branaplam 56 mg | Overall
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/5 | 4/21 | 4/26
Other Adverse Events (participants affected / at risk) | 2/5 | 15/21 | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Branaplam 56 mg (N=21) | Overall (N=26)
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 2
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Branaplam 56 mg (N=21) | Overall (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 5
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Puncture site pain (General disorders) | 0 | 3 | 3
COVID-19 (Infections and infestations) | 1 | 2 | 3
Cystitis (Infections and infestations) | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Balance disorder (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 2 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 2 | 3
Polyneuropathy (Nervous system disorders) | 0 | 3 | 3
Delusional disorder, persecutory type (Psychiatric disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT05111249/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT05111249/SAP_001.pdf